CLINICAL TRIAL: NCT03115567
Title: A Randomized Phase II Study of Topical Steroids as Preemptive Therapy for Epidermal Growth Factor Receptor Inhibitor-Induced Papulopustular Eruption
Brief Title: A Study of Topical Steroids as Preemptive Therapy for EGFR Inhibitor-Induced Papulopustular Eruption
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment accrual
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Nam Choi, MD, Chief of Oncodermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JNC06142016
Record Dates: First submitted 2017-02-15; First posted 2017-04-14 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Acneiform Rash; Papulopustular Eruption
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in Control group will be instructed to follow a daily moisturizer and sunscreen regimen. Erlotinib, cetuximab, panitumumab, or afatinib will be administered as standard of care treatment.
- Triamcinolone (Experimental): Patients in the Triamcinolone group will be applying Triamcinolone 0.1% cream daily to their face, chest, and upper back, in addition to adhering to the same daily moisturizer and sunscreen regimen of the Control group. Erlotinib, cetuximab, panitumumab, or afatinib will be administered concomitantly as standard of care treatment.
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — 6 weeks of twice daily application of 0.1% triamcinolone cream to the face, chest, and back.
  Arms: Triamcinolone

SUMMARY:
This randomized, controlled, phase II clinical study is designed to assess the efficacy of preemptive treatment with topical steroids in preventing the papulopustular eruption induced by epidermal growth factor receptor inhibitor (EGFRI) treatment in cancer patients. Participants will be followed up for 6 weeks of twice daily application of triamcinolone cream to the face, chest, and back.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed cancer diagnosis for which EGFRI treatment is indicated
* Initiation of topical steroids or control treatment within 3 days of initiation of cetuximab, erlotinib, panitumumab, or afatinib
* Patients must be age ≥ 18 years.
* Life expectancy of greater than 6 weeks
* Patient able to use topical medications reliably and complete questionnaires with assistance if needed
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

* Patients who have used systemic or topical steroids within 7 days of trial registration, or start systemic or topical steroids for reasons unrelated to trial during the 6-week follow up period
* Patients who have used antibiotics within 7 days of trial registration, or start antibiotics for other conditions during the 6-week follow up period
* History of allergic reactions to topical steroids
* Patients with any rash at the time of study registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients using any other topical medications in the treatment areas (face, chest, or back).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Choi, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacouture ME, Maitland ML, Segaert S, Setser A, Baran R, Fox LP, Epstein JB, Barasch A, Einhorn L, Wagner L, West DP, Rapoport BL, Kris MG, Basch E, Eaby B, Kurtin S, Olsen EA, Chen A, Dancey JE, Trotti A. A proposed EGFR inhibitor dermatologic adverse event-specific grading scale from the MASCC skin toxicity study group. Support Care Cancer. 2010 Apr;18(4):509-22. doi: 10.1007/s00520-009-0744-x. Epub 2010 Feb 10. PMID 20145956

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Triamcinolone
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Triamcinolone | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 7 | 0 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: % of Participants With Grade 2 Rash or Higher
Description: To assess the difference in percentage of participants who develop a grade 2 or greater rash in the control group as compared to the case group of preemptive treatment with topical steroids (triamcinolone 0.1% cream for application to face, chest and back) when administered concomitantly for 6 weeks with erlotinib, cetuximab, panitumumab, or afatinib to prevent papulopustular eruptions.
Time Frame: 6 weeks
Population: Analysis completed on N=6 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Triamcinolone
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

2. Secondary Outcome: Change in Quality of Life Using FACT-EGFRI 18 Quality of Life Assessment
Description: To assess the difference in change in quality-of-life due to rash at Visit 4 from Visit 1 between the two treatment groups. FACT-EGFRI 18 is an 18-question assessment for cancer patients undergoing EGFR treatment. The scoring range is 0-72, with 72 indicating more severe functional impact.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Triamcinolone
Number analyzed (Participants) | 4 | 7
score on a scale | 14.25 [6 to 24] | 4.57 [-2 to 14]

3. Secondary Outcome: Number of Participants in the Treatment and Control Group Who Adhere to Their Chemotherapy Regimen Determined by Whether Patients Discontinue Their Chemotherapy Regimen or Continue Their Full Course of Treatment
Description: This measure is to determine if the control group discontinues their chemotherapy regimen more often than the treatment group
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Triamcinolone
Number analyzed (Participants) | 3 | 3
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 3 years and 3 months
Arm/Group | Control | Triamcinolone
All-Cause Mortality (participants affected / at risk) | 3/7 | 4/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03115567/Prot_SAP_000.pdf